CLINICAL TRIAL: NCT02399501
Title: Sonohysterography and 3D Ultrasonography Versus Diagnostic Hysteroscopy in Assessment of Uterine Factor in Cases of Female Infertility
Brief Title: Sonohysterography , 3D Ultrasonography and Hysteroscopy in Assessment of Uterine Factor in Cases of Female Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 132
Record Dates: First submitted 2015-03-05; First posted 2015-03-26 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Infertility
Keywords: 2D ultrasound; 3D ultrasound; sonohysterography; hysteroscopy; Uterine factor of infertility
MeSH Terms: conditions — Infertility | interventions — Hysteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- uterine lesion ultrasound, hysteroscopy (Experimental): evaluation of female with proved uterine lesion by two dimensional ultrasound, three dimensional ultrasound, saline sonohysterography and hysteroscopy
  Interventions: Procedure: hysteroscopy; Device: two dimensional ultrasound; Device: saline sonohysterography; Device: three dimensional ultrasound

INTERVENTIONS:
Procedure: hysteroscopy — Hysteroscopy is done under general anesthesia. The hysteroscopy used is rigid continuous flow diagnostic hysteroscopy (Tuttligen, Karl Storz, Germany). It has a 30º panoramic optic which is 4 mm in diameter and the diagnostic continuous flow outer sheath is 6.5 mm in diameter.
Device: two dimensional ultrasound — Examination is performed after emptying of the bladder in dorsal lithotomy position .The probe is introduced into the posterior fornix of the vagina, then the following structures are examined, the uterus for site, size and mobility, the myometrium for fibroids and adenomyosis, the endometrium for uniformity, polyps, submucous fibroids and intrauterine adhesions, the cervix for nabothian follicles and polyps, the adenexa and ovaries for site, size, mobility, follicles, cysts and corpus luteum
  Other Names: (Sonoace 5000)
Device: saline sonohysterography — sterile speculum is introduced and the vagina and cervix is cleaned with povidone iodine 10%. Cook ET (embryo transfer) catheter is used. . After introduction of the catheter into the cervix, a twenty milliliter syringe which will be prefilled with the distending media (saline) then fitted to the catheter. The speculum is removed and endovaginal probe is introduced in the posterior vaginal fornix
  Other Names: (Sonoace 5000)
Device: three dimensional ultrasound — The uterus is visualized in the longitudinal plane, the ultrasound probe is kept steady and the patient is asked to lie still on the examination bed. The volume mode is switched on. Three D volume is generated by the automatic rotation of the mechanical transducer through 360º. The acquired volume is in the shape of a transacted cone with a depth of 4.3 - 8.6 cm and a vertical angle α = 90º. Using the medium line density, the typical acquisition time is a round 10 seconds
  Other Names: (Medison, Voulson 530 D-MT ultrasound machine)

SUMMARY:
Prospective comparative study including 100 infertile patients with suspected uterine lesion. 2D ultrasound, sonohysterography , 3D ultrasound and hysteroscopy will be done to evaluate uterine cavity.

DETAILED DESCRIPTION:
All patients will be examined by 2D transvaginal ultrasound using a 6.5 MHz probe (Sonoace 5000, Medison Co. Ltd, korea). Examination is performed after emptying of the bladder in dorsal lithotomy position.

Three dimensional ultrasound will be performed using Medison, Voulson 530 D-MT ultrasound machine (Medison Co. Ltd, Korea). The uterus is visualized in the longitudinal plane, the ultrasound probe is kept steady and the patient is asked to lie still on the examination bed.

Sonohysterography will be done after introduction of the catheter into the cervix, a twenty milliliter syringe which is prefilled with the distending media (saline) is then fitted to the catheter. The speculum is removed and endovaginal probe is introduced in the posterior vaginal fornix. The uterus is then visualized in the longitudinal plane to demonstrate the endometrial cavity and the catheter. Once this is possible, sterile saline is slowly injected through the catheter into the uterine cavity; up to ten milliliter of saline is usually enough for the procedure.

Hysteroscopy will be done under general anesthesia. The hysteroscopy is rigid continuous flow diagnostic hysteroscopy . It has a 30º panoramic optic which is 4 mm in diameter and the diagnostic continuous flow outer sheath is 6.5 mm in diameter.

ELIGIBILITY:
Inclusion Criteria:

* Suspected uterine factor of infertility

Exclusion Criteria:

* tubal, ovarian or male factor of infertility

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
detection of uterine lesion | at time of hystroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Ahmed Maged, Cairo, Egypt